CLINICAL TRIAL: NCT05275647
Title: Therapeutic Efficacy and Safety of Low Energy Shock Wave (LESW) Plus Botulinum Toxin A Instillation in Treatment of Patients With Interstitial Cystitis Refractory to Conventional Therapy - A Clinical and Immunohistochemistry Study
Brief Title: Efficacy and Safety of Low Energy Shock Wave Plus BotulinumToxin A in Treating Patients With Interstitial Cystitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); Hualien Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Hann-Chorng Kuo, M.D., Chairman, Department of Urology, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 110-078-A
Record Dates: First submitted 2022-01-13; First posted 2022-03-11 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Interstitial Cystitis
Keywords: Low energy shock wave; interstitial cystitis; botulinum toxin A; urothelium
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Botulinum Toxins, Type A; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized, placebo-controlled physician initiated study enrolled patients with refractory IC/BPS.
Who Masked: Participant, Investigator
Masking Description: Participants and investigator are blinded to the treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group : BoNT-A 100 U in Normal saline (Experimental): BOTOX 100U in normal saline (BoNT-A/NS) 30ml in single intravesical instillation
  Interventions: Drug: BOTOX 100U in normal saline
- Placebo group : Normal saline (Placebo Comparator): Normal saline (N/S) 30ml in single intravesical instillation
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: BOTOX 100U in normal saline — LESW with 3000 shocks, frequency of 3 pulses per second, and maximum total energy flow density 0.25 mJ/mm2 , and followed by intravesical BoNT-A 100U instillation in 30ml normal saline retained in the bladder for 2 hours, every one week for 4 times.
  Other Names: BOTOX
  Arms: Treatment group : BoNT-A 100 U in Normal saline
Drug: Normal saline — LESW treatment with 3000 shocks, frequency of 3 pulses per second, and maximum total energy flow density 0.25 mJ/mm2 , and followed by intravesical instillation of 30ml normal saline retained in the bladder for 2 hours after LESW application, every one week for 4 times.
  Other Names: Saline
  Arms: Placebo group : Normal saline

SUMMARY:
Low energy shock wave (LESW) is known to facilitate tissue regeneration with analgesic and anti-inflammatory effects. LESW treatment has been demonstrated effective in treatment of nonbacterial prostatitis and chronic pelvic pain syndrome. LESW reduced pain behavior and down-regulated the NGF expression, suppressed bladder overactivity by decreasing inflammation, IL-6 and COX2 expression and NGF expression. Previous rat interstitial cystitis (IC) models have shown LESW could increase urothelial permeability, facilitate intravesical botulinum toxin A (BoNT-A) delivery and block acetic acid induced hyperactive bladder, suggesting LESW might be a potential therapeutic candidate for relieving bladder inflammatory conditions and overactivity. A double-blind, randomized, placebo-controlled physician-initiated study revealed LESW treatment was associated with a statistically significant decrease in O'Leary-Saint Symptom Score and visual analog scale of pain in patients with interstitial cystitis/bladder pain syndrome (IC/BPS), but the improvement was not superior to the sham LESW treatment. Previous studies found the urothelial dysfunction and deficits of cell differentiation are fundamental pathophysiology of IC/BPS. Through intravesical platelet-rich plasma injections, the chronic inflammation in IC/BPS bladders could be reduced and improved cell differentiation of urothelium. Botox injection or liposome encapsulated Botox could also inhibit inflammation and improve IC/BPS symptoms. However, the Botox injection needs anesthesia and certain complications might occur. There is no study to test if LESW plus Botox intravesical instillation could improve bladder inflammation and relieve IC/BPS symptoms. This study aims to investigate the therapeutic efficacy and safety of concomitant LESW plus intravesical BoNT-A instillation for IC/BPS refractory to conventional treatments.

DETAILED DESCRIPTION:
Interstitial cystitis/ bladder pain syndrome (IC/BPS) is a bladder disorder with unknown etiology and difficult treatment. Novel treatments have been searched to adequately improved symptoms. Low energy shock wave (LESW) increased urothelial permeability, facilitated intravesical botulinum toxin A (BoNT-A) delivery and blocked acetic acid induced hyperactive bladder. Rats that received BoNT-A plus LESW showed a significantly reduced response (48.6% decreased intercontractile interval) to acetic acid instillation without compromising voiding function. Rats pre-treated with BoNT-A plus LESW showed a decreased inflammatory reaction (p <0.05), and decreased expressions of SNAP-23 (p < 0.05), SNAP-25 (p = 0.061) and COX-2 (p < 0.05) compared with the control group. These results support LESW as a promising method to deliver BoNT-A across urothelium without the need for injection. LESW is known to facilitate tissue regeneration with analgesic and anti-inflammatory effects. LESW treatment reduced pain behavior and down-regulated the NGF expression (33.3%, P < 0.05) on day 4 and IL-6 (40.9%, P < 0.05). LESW treatment suppressed bladder overactivity (intercontractile interval 77.8% increase, P < 0.05) by decreasing inflammation and COX2 (38.6%, P < 0.05) expression and NGF expression (25.2%, P = 0.0812). Previous study revealed that LESW might be a potential candidate for relieving bladder inflammatory conditions and overactivity. Recent clinical trial also revealed that Intravesical instillation of BoNT-A and LESW is a safe and effective method for the treatment of refractory overactive bladder with a durable response for 2 months. A double-blind, randomized, placebo-controlled physician-initiated study enrolled 54 patients with IC/BPS. The patients were assigned to LESW or placebo. At 4 weeks post-treatment, both groups were associated with a statistically significant decrease in OSS and VAS pain scale. A significantly higher proportion of patients on LESW responded as improved in the VAS ≥ 3 vs placebo (P = 0.035). At 12 weeks post-treatment, improvement in the VAS ≥ 3 was 57.1% vs 19.0% (LESW vs placebo; P = 0.011). No significant adverse events were found in either group. This study aims to investigate the therapeutic efficacy and safety of concomitant LESW plus intravesical BoNT-A instillation for IC/BPS patients refractory to conventional treatments.

Materials and Methods

Eligible participants of either gender with IC/BPS refractory to at least two treatments will be enrolled to this study. Participants are randomly allocated to receive either treatment in 1:1 ratio according to the permuted block randomization code as the following:

(A) LESW treatment with 3000 shocks, and followed by intravesical instillation of 30ml normal saline. (placebo group)

(B) LESW with 3000 shocks, and followed by intravesical BoNT-A 100U instillation. (treatment group)

Urine samples will be collected for urinary protein and biomarkers analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with age of 20 years old or above
2. Patients with symptoms of frequency, urgency, and bladder pain at full bladder for more than 6 months.
3. Proven to have glomerulations (at least grade 1) by cystoscopic hydrodistention under anesthesia in recent 1 year
4. Free of active urinary tract infection
5. Free of bladder outlet obstruction on enrolment
6. Free of overt neurogenic bladder dysfunction and limitation of ambulation.
7. Patient or his/her legally acceptable representative agrees to sign the written informed consent form

Exclusion Criteria:

1. Patient's lower urinary tract symptoms can be effectively treated by conventional therapy
2. Patient or his/her legally acceptable representative cannot sign the written informed consent form
3. Patient cannot complete the consecutive 3- day voiding diary on the visiting day
4. Patient had been treated for overactive bladder by enterocystoplasty
5. Patients with severe cardiopulmonary disease and such as congestive heart failure, arrhythmia, poorly controlled hypertension, not able to receive regular follow-up
6. Patient has bladder outlet obstruction on enrollment
7. Patients has post-void residual >250ml
8. Patients with uncontrolled confirmed diagnosis of acute urinary tract infection
9. Patients have laboratory abnormalities at screening including: ALT> 3 x upper limit of normal range, AST> 3 x upper limit of normal range; Patients have abnormal serum creatinine level > 2 x upper limit of normal range
10. Patient has coagulation disorder
11. Female patients who is pregnant, lactating, or with child-bearing potential without contraception.
12. Patients with any other serious disease considered by the investigator not in the condition to enter the trial
13. Patient had received intravesical hyaluronic acid insillation treatment for IC within recent 6 months before enrolment
14. Patient had received intravesical onabotulinumtoxinA treatment for IC within recent 12 months before enrolment
15. Patients participated investigational drug trial within 1 month before entering this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-05-18 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
O'Leary-Sant Symptom Score | from baseline to 3 month after the treatment day
  Change of the O'Leary-Sant symptom score (including Interstitial Cystitis Symptom Index from 0 to 10 points and Interstitial Cystitis Problem Index, from 0 to 20 points; a higher score indicates a worse symptom severity)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | from baseline to 3 month after the treatment day
  Local or systemic adverse events such as hematuria, miction pain, difficult urination, or any systemic symptoms such as fever, general weakness, dyspnea, etc.)

SECONDARY OUTCOMES:
Global response assessment (GRA) | 1 month after the treatment day
  Global response assessment (GRA) of satisfaction by the patient (categorized into -3, -2, -1, 0, 1, 2, 3 units of scale, indicating markedly worse to markedly improved) at 1 month after the treatment day.
  An improvement of GRA by 2 units of scale at 1 month is considered effective.
Visual analog score (VAS) for pain | from baseline to 1 month and 3 months after the first treatment day
  Net change of the Visual analog score (VAS) for pain (from 0 to 10 units of scale, indicating no pain (0) to severe pain (10))
Functional bladder capacity | from baseline to 1 month and 3 months after the first treatment day
  Net change of functional bladder capacity (FBC, in milliliter)
Voiding frequency per day | from baseline to 1 month and 3 months after the first treatment day
  Net change of voiding frequency at daytime and voiding frequency at night time as record in 3-day voiding diary
maximum flow rate | from baseline to 1 month after the first treatment day
  Net changes of the maximum flow rate (Qmax, in milliliter/second)
voided volume | from baseline to 1 month after the first treatment day
  Net changes of the voided volume (in milliliter)
Pos-tvoid residual volume (PVR) | from baseline to 1 month after the first treatment day
  Net changes of the PVR (in milliliter)
urinary nerve growth factor (NGF) | from baseline to 1 month and 3 months after the first treatment day
  Changes of urinary NGF level in urine (in nanogram/milliliter)
urinary brain derived neurotrophic factor (BDNF) | from baseline to 1 month and 3 months after the first treatment day
  Changes of urinary BDNF (in nanogram/milliliter)
Inflammatory cytokine IL-2 level | from baseline to 1 month and 3 months after the first treatment day
  Changes of cytokine IL-2 level (in nanogram/milliliter)
Inflammatory cytokines IL-6 level | from baseline to 1 month and 3 months after the first treatment day
  Changes of cytokines IL-6 level (in nanogram/milliliter)
Inflammatory cytokine IL-8 level | from baseline to 1 month and 3 months after the first treatment day
  Changes of cytokine IL-8 level (in nanogram/milliliter)
Inflammatory cytokine IL-1 beta level | from baseline to 1 month and 3 months after the first treatment day
  Changes of cytokine IL-1 beta level (in nanogram/milliliter)
Safety outcome (Local and systemic adverse events) | from baseline to 1 month and 3 months after the first treatment day
  Any adverse events occurring after treatment, including hematuria, micturition pain, difficulty in urination, urinary tract infection, or systemic symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Hann-Chorng Kuo, M.D., Principal Investigator — Department of Urology, Buddhist TzuChi General Hospital
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No